CLINICAL TRIAL: NCT03236233
Title: A Randomised, Single-blind, Placebo-controlled, Dose-escalation Study to Assess the Safety and Tolerability of Single and Repeat, Inhaled Doses of PC786 in Healthy Subjects Combined With a Randomised, Single-blind, Placebo-controlled, Parallel Group to Assess the Safety and Tolerability of a Single Dose of Inhaled PC786 in Subjects With Mild Asthma
Brief Title: A Study to Investigate the Safety and Tolerability of Single and Repeat Doses of PC786
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC_RSV_001; 2016-000934-22 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-08-01 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — PC-786

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose - healthy subjects (Experimental)
  Interventions: Drug: PC786 - Single doses; Drug: Placebo - Single doses
- Repeat dose - healthy subjects (Experimental)
  Interventions: Drug: PC786 - Repeat doses; Drug: Placebo - Repeat doses
- Single dose - subjects with asthma (Experimental)
  Interventions: Drug: PC786 - Single doses; Drug: Placebo - Single doses

INTERVENTIONS:
Drug: PC786 - Single doses — Safety and tolerability of single doses
  Arms: Single dose - healthy subjects; Single dose - subjects with asthma
Drug: Placebo - Single doses — Safety and tolerability of single doses
  Arms: Single dose - healthy subjects; Single dose - subjects with asthma
Drug: PC786 - Repeat doses — Safety and tolerability of repeat doses
  Arms: Repeat dose - healthy subjects
Drug: Placebo - Repeat doses — Safety and tolerability of repeat doses
  Arms: Repeat dose - healthy subjects

SUMMARY:
This study investigates the safety, tolerability and pharmacokinetics of single and repeat doses of PC786.

ELIGIBILITY:
Inclusion Criteria:

All subjects (Cohorts 1, 2, 3 & 4)

* Must be male or female, aged between 18 and 65 years inclusive (at the time of consent) who fit one of the following criteria: women of childbearing potential who are willing and able to use contraception from screening until 30 days after receipt of the final dose; Women of non-childbearing potential defined as being amenorrhoeic or have been permanently sterilised; Men who are willing and able to use contraception from the time of the first dose, until 90 days after receipt of the final dose of study medication.
* Females must have a negative serum β human chorionic gonadotropin (β-hCG) test at screening and a negative urinary pregnancy test at Day -1.
* Subject must be willing and able to adhere to the restrictions and prohibitions required by this protocol.
* Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose and requirements of the study and that they are willing to participate.
* Body weight ≥ 50 kg and body mass index (BMI) within the range 18 - 30 kg/m2 (inclusive).
* Average QTcF <450 msec at screening and pre-dose.
* Vital signs assessments within normal ranges at screening and pre-dose.

Healthy Subjects (Cohorts 1, 2 & 3)

* Healthy as determined by a physician based on a full medical examination including medical history, physical examination and laboratory tests performed at screening and pre-dose.
* Spirometry readings (FEV1 and FVC) to be ≥ 80% of predicted value and FEV1/FVC ratio > 0.7 at screening

Subjects with Asthma (Cohort 4)

* Documented diagnosis of asthma, first diagnosed at least 12 months prior to the screening visit.
* Subject must demonstrate a PC20 methacholine ≤ 8 mg/mL at the screening visit.
* Have an FEV1 >60% of predicted normal value at least 6 h after the last use of a short acting β-agonist (SABA).
* Have stable asthma based on physician assessment at screening and prior to randomisation
* Subject must be otherwise healthy on the basis of a full medical examination including medical history, physical examination and laboratory tests performed at screening.

Exclusion Criteria:

All subjects (Cohorts 1, 2, 3 & 4)

* Any acute illness.
* Upper or lower respiratory tract infection within 4 weeks of the screening visit or randomisation.
* Use of prescription medications within 14 days of the Screening visit
* Are taking over the counter medications other than vitamins or multivitamins and herbal medication, within 14 days prior to Screening
* History of regular alcohol consumption within 6 months of the study of an average weekly intake of >21 units for males, or >14 units for females
* Definite or suspected history of drug or alcohol abuse within the previous 5 years.
* A smoker (regular or irregular), or has smoked or used nicotine-containing products (including e-cigarettes) within the 6 months prior to screening
* A positive test for HIV-1 & -2 antibodies at screening.
* A positive pre-study hepatitis B surface antigen or positive hepatitis C antibody result at screening.
* Positive test for alcohol, smoking or drugs of abuse, at screening or pre-dose
* Received an experimental drug or used an experimental medical device within 3 months before the first dose of the study drug is scheduled.
* Allergy to any of the active or inactive ingredients in the study medication.
* History of drug, or other allergy that would contraindicate participation.
* Donation of blood in excess of 500 mL within a 3 month period prior to dosing
* Mentally or legally incapacitated.
* An employee of the Sponsor or contract research organisation (CRO), or a relative of an employee of the Sponsor or CRO.
* Unable or unwilling to undergo multiple venepuncture procedures
* Pregnant or lactating female
* Any other reason that the Investigator considers makes the subject unsuitable to participate.

Healthy Subjects (Cohorts 1, 2 & 3)

* Any chronic illness or clinically relevant abnormality identified on the screening medical assessment, laboratory tests or ECG

Subjects with Asthma (Cohort 4)

* Has ever had an episode of life-threatening asthma defined as respiratory arrest, intubation for asthma, or ICU admission for asthma.
* Presence of clinically significant diseases other than asthma, hyper-responsive airways, seasonal allergic rhinitis or atopic diseases
* Has experienced an acute asthma exacerbation in the 12 months prior to screening requiring hospitalisation or accident and emergency treatment or management with systemic or injectable steroids.
* Has uncontrolled, or moderate to severe asthma based on PI assessment and/or use of prohibited medications, or has required treatment with these therapies in the previous 12 weeks.
* History or presence of any known conditions contraindicated for methacholine challenge

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting one or more treatment-emergent adverse events (TEAE) | Baseline up to Week 12
Number of participants who discontinue due to an adverse event (AE) | Baseline up to Week 12
Number of participants who meet the markedly abnormal criteria for safety 12-lead ECG assessment at least once post dose | Baseline up to Week 12
Number of participants who meet the markedly abnormal criteria for vital signs assessment at least once post dose | Baseline up to Week 12
Number of participants who meet the markedly abnormal criteria for safety laboratory assessments at least once once post dose | Baseline up to Week 12
Number of participants who meet the markedly abnormal criteria for safety spirometry assessment (FEV1 & FVC - measured together) at least once once post dose | Baseline up to Week 12

SECONDARY OUTCOMES:
Plasma concentration of PC786 | Day 1: Pre-dose and at multiple time points (up to 10 days) post final dose
  Blood levels of PC786 measured after dosing
Mucosal lining fluid concentration of PC786 | Cohort 1 - Day 1 = 3 samples; Day 2 = 2 samples; Day 3 = 1 sample. Cohorts 2 & 3 - Day 1 = 2 samples; Day 6 = 1 sample; Day 7 = 3 samples; Day 8 = 2 samples; Days 9 & 10 - 1 sample
  PC786 concentration data in mucosal lining fluid measured after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J Boyce, MBChB, MD, Principal Investigator — cro
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom